CLINICAL TRIAL: NCT06018779
Title: Effectiveness of Cryo Plus Ultrasound Therapy Versus Diathermy in Combination With High-intensity Laser Therapy for Pain Relief in Footballers With Muscle Injuries: a Prospective Study
Brief Title: Effectiveness of Physical Therapy for Pain Relief in Footballers With Muscle Injuries: a Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof.ssa Giulia Letizia Mauro, Professor, University of Palermo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MFR0032023
Record Dates: First submitted 2023-08-21; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Athletic Injuries; Physical Therapies
MeSH Terms: conditions — Athletic Injuries | interventions — Diathermy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Group A will include patients who will receive a rehabilitation treatment consisting of: cryo-ultrasound therapy and high-intensity laser therapy
  Interventions: Other: Cryoultrasound therapy plus high-intensity laser therapy
- Group B (Placebo Comparator): Group B will include patients who will receive a rehabilitation treatment consisting of: cryo-ultrasound therapy and diathermy
  Interventions: Other: diathermy plus high-intensity laser therapy

INTERVENTIONS:
Other: Cryoultrasound therapy plus high-intensity laser therapy — Group A received a daily rehabilitation treatment lasting 10 sessions for 10 consecutive sessions, consisting of high-intensity laser therapy and cryo-sound therapy.
  Arms: Group A
Other: diathermy plus high-intensity laser therapy — Group B received a daily rehabilitation treatment lasting 10 sessions for 10 consecutive sessions, consisting of high-intensity laser therapy and diathermy.
  Arms: Group B

SUMMARY:
The objective of this study was to evaluate the efficacy of cryoultrasound therapy versus diathermy in combination with high-intensity laser therapy for pain relief in male professional soccer players with muscle injuries. The main questions it intends to answer are:

• Is this combination of treatments effective in these patients in terms of pain relief?

Participants will receive a rehabilitation treatment consisting of cryo-ultrasound therapy and high intensity laser. Researchers will compare the group of participants, called the treatment group, with a control group to see if:

• Is the combined treatment of cryoultrasound therapy and high intensity laser more effective in these patients than the combination of diathermy and high intensity laser?

ELIGIBILITY:
Inclusion Criteria:

* age 18-21 years;
* professional footballer in a competitive club;
* presence of a grade III A muscle lesion, according to the Mueller-Wohlfart classification, confirmed by ultrasound examination and occurring during sports activity at least 5 days before inclusion in the present study;
* no previous muscle injuries in the last 6 months;
* signature of the written informed consent for participating in the study.

Exclusion Criteria:

* previous muscle injuries or bone fractures of the lower limbs in the last 6 months;
* knee instability due to previous rupture of knee ligaments;
* active neoplastic or infectious diseases;
* congenital anomalies of the lower limbs.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
entity of the pain | 2 weeks
  numerical rating scale; the total score ranges from 0 to 10, with higher scores indicating more pain.

SECONDARY OUTCOMES:
size of the muscle tear | 2 weeks
  measurement in centimeters by ultrasound.
frequency of relapses | 3 months after the injury
  number of relapses
return to play | 3 months after the injury
  number of days

CONTACTS AND LOCATIONS:
Locations (1):
- Functional Recovery and Rehabilitation Unit of the A.O.U.P. Paolo Giaccone, Palermo, Italy